CLINICAL TRIAL: NCT04739098
Title: Initial Manifestations of Congestive Heart Failure in Patients With Non-ST-segment Elevation Acute Coronary Syndrome
Brief Title: Initial Manifestations of Congestive Heart Failure in Patients With NSTEACS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Medical Research Center for Therapy and Preventive Medicine (Other Government)
Collaborators: Moscow City Hospital named after A.K. Eramishantsev (Other Government)
Responsible Party: Sponsor
Other Study IDs: 7
Record Dates: First submitted 2021-02-01; First posted 2021-02-04 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Acute Heart Failure, Non-ST-segment Elevation Acute Coronary Syndrome
Keywords: acute heart failure, congestive heart failure, non-ST-segment elevation acute coronary syndrome, lung ultrasound, vena cava inferior ultrasound
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute heart failure (HF) is a common complication of acute coronary syndrome (ACS) associated with poor prognosis. Diagnosis of congestive HF in patients with initial, non-severe symptoms and signs may be challenging and early stages of this complication may be missed. To assess severity of HF in patients with ACS Killip classification is widely used but it does not take into account mild manifestations of HF. Thus, patients without rales in the lungs and/or S3 will be labelled as Killip class 1. The aim of this study is to determine the frequency, risk factors, abilities for early diagnosis using routine medical evaluation and clinical significance of subclinical and mildly symptomatic congestive HF in patients with ACS without persistent ST-segment elevation (NSTEACS).

The study will include 200 patients with NSTEACS without history of severe HF and overt signs of congestion at presentation. Presence and severity of dyspnea (according to Likert ans Visual analog scales), physical signs of heart failure (respiratory rate, distention of jugular veins, S3), peripheral oxygen saturation by pulse oximetry, heart rate and signs of ischemia on ECG, signs of congestion according to lung and vena cava inferior ultrasound and chest X-Ray/CT as well as levels of NT-proBNP, hsTn, CRP and FABP at presentation will be evaluated. Presence and severity of dyspnea, physical signs of heart failure, oxygen saturation, heart rate and signs of ischemia on ECG, lung and vena cava inferior ultrasound will be re-assessed after 6, 12 and 24 hours. During hospitalization occurrence or worsening of clinical HF. Clinical events will be followed up to 12 months after hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized to the cardiac intensive care unit with ACS without persistent ST-segment elevation
* Signed informed consent

Exclusion Criteria:

* ACS with persistent ST-segment elevation
* High probability of absence of ACS
* Congestive rales in the base of lungs, cardiac asthma, pulmonary edema, cardiogenic shock, obvious edema, anasarca
* History of severe chronic heart failure (III-IV NYHA class, obvious edema, anasarca)
* Continuous use of loop diuretics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ACS without persistent ST-segment elevation without history of severe HF and clinical signs of congestion at presentation
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-01-30 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2024-08-28 (Estimated)

PRIMARY OUTCOMES:
Worsening of HF from enrollment to 24 hours | from enrollment up to 24 hours
  Worsening of HF is stated if at least one of following is present
  1. ≥1 point increase of dyspnea according to 5-point Likert score: 1=not short of breath, 2=mildly short of breath, 3=moderately short of breath, 4=severely short of breath, 5=very severely short of breath.
  2. Appearance/increase of jugular vein distension (if starting to be seen in patients lying horizontally or increasing degree of head of bed elevation for its disappearance).
  3. Appearance of S3 gallop.
  4. Appearance of congestive rales in the lungs.
  5. Appearance of peripheral oedema related to HF.
  6. Intravenous administration of diuretics/vasodilators due to clinical deterioration of HF.

SECONDARY OUTCOMES:
Changes severity of congestion according to lung and vena cava inferior ultrasound from enrollment to 24 hours after initial assessment at presentation | from enrollment up to 24 hours
Composite of death, (re)myocardial infarction, stroke or hospitalisation for 12 months | up to 12 months
Composite of death, (re)infarction, stroke or worsening of HF from enrollment to discharge from the hospital | from admission to discharge or death during reference hospitalization, assessed up to 90 days
  Worsening of HF is stated if at least one of following is present
  1. Appearance of congestive rales in the lungs.
  2. Appearance of peripheral oedema related to HF.
  3. Intravenous administration of diuretics/vasodilators due to clinical deterioration of HF.

CONTACTS AND LOCATIONS:
Locations (1):
- National Medical Research Center for Therapy and Preventive Medicine of the Ministry of Health of the Russian Federation and City clinical hospital named after A. K. Eramishantsev, Moscow, Russia, 129327, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No